CLINICAL TRIAL: NCT06071585
Title: Monocentric Retrospective Observational Study for Validation of Meta-analysis of the Metatrascryptome and Transcriptome of Eosynophyl Esophagitis (EoE TaMMA)
Brief Title: Monocentric Retrospective Observational Study for Validation of Meta-analysis of the Metatrascryptome and Transcriptome of Eosynophyl Esophagitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Director of Gastroenterology and Endoscopy Unit, IRCCS San Raffaele
Other Study IDs: EoE TaMMA
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with Eosinophilic esophagitis (EoE)
  Interventions: Other: Formalin-fixed Paraffin-embedded (FFPE) tissue samples analysis
- patients with gastroesophageal reflux disease (GERD)
  Interventions: Other: Formalin-fixed Paraffin-embedded (FFPE) tissue samples analysis
- controls (patients without EoE e GERD)
  Interventions: Other: Formalin-fixed Paraffin-embedded (FFPE) tissue samples analysis

INTERVENTIONS:
Other: Formalin-fixed Paraffin-embedded (FFPE) tissue samples analysis — We will stain and analyze EoE, GERD, and controls Formalin-fixed paraffin-embedded (FFPE) tissue samples already stored in the pathological laboratory of OSR.

SUMMARY:
This is a retrospective monocentric observational study involving patients with Eosinophilic esophagitis (EoE), gastroesophageal reflux disease (GERD), and controls (patients without EoE and GERD). To validate the EoE-related markers obtained with the EoE TaMMA web app (such as CCL26, TBX5, NOX4, FGF7, CXCL14, ADAMTS5, PDGFRA, CXCL12, ACVRL1, POSTN, and LTBP4), we will stain and analyze EoE, GERD, and controls Formalin-fixed paraffin-embedded (FFPE) tissue samples already stored in the pathological laboratory of OSR. For this reason, this project will be accomplished thanks to the collaboration with prof.

Doglioni's team at OSR.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a chronic esophageal inflammatory disease, primarily activated by food antigens, with the concomitant accumulation of eosinophils within the esophageal mucosal layer where the Th2-response-specific interleukin (IL) 5 and IL13 play a key role during its pathogenesis. EoE positions as an uncommon disease, with a suggested genetic basis and a 3:1 male preponderance. Its incidence rate varies between 0.1 and 1.2 cases per 10,0009 and increases annually. EoE symptoms include difficulty with eating, failure to thrive, vomiting, chest and/or abdominal pain, dysphagia, and food impaction, histologically associated with esophageal linear furrows with loss of vascularity, mucosal rings, a small-caliber lumen, strictures, mucosal exudates, and, less commonly, polyps and ulcerations. The currently adopted therapies are mainly based on proton pump inhibition, topical administration of glucocorticoids, and changes in dietary habits. However, in most patients, eosinophilic esophagitis remains a chronic disease, and if treatment is stopped, inflammation ensues and symptoms recur. This may hamper the quality of life, including vitality and general health scores, and complications may develop. Therefore, the complete comprehension of the mechanisms occurring during EoE pathogenesis remains of paramount importance to implementing and improving the therapeutic lines of intervention, ameliorating the overall patients' wellness.

A straightforward and facilitated EoE clinical diagnosis is still missing, since EoE provokes in patients symptoms overlapping with other disease manifestations, such as gastroesophageal reflux disease (GERD), eosinophilic gastrointestinal disease, and achalasia. Along with the mucosal immunity alterations, the epithelial barrier function impairment does remain a hallmark of EoE, in terms of both increased permeability and antigen sensing and EoE TaMMA .

Indeed, at the mucosal level, EoE is featured by a striking pattern of dilated interepithelial spaces, with down-regulation of proteins associated with barrier function and adhesion molecules, in turn, modulated via an IL13-dependent mechanism. As a consequence, altered epithelial permeability can lead to a permissive environment that enhances antigen presentation, which in turn leads to persistent chronic inflammation.

Despite some anatomical and molecular characterizations employed as a kind of gold standard for the definition of the EoE pathogenesis, a meta-analysis of the molecular studies may improve the understanding of the physiopathology of the disease and define molecular markers helpful for a straightforward diagnosis of EoE has not been performed yet. We recently developed and released the Inflammatory Bowel Disease (IBD) Transcriptome and Metatranscriptome Meta-Analysis web app (IBD TaMMA, https://ibd-meta-analysis.herokuapp.com/), a complete survey of all public data sets generated for IBD-related studies. TaMMA has contributed to the field of omics data meta-analysis by providing an open source framework that will enable the community to easily access, query, and 'play' with the data through a user-friendly web application and offering an unprecedented opportunity to define new hypotheses and insights for better understanding the pathogenesis of IBD.

Considering the utility that IBD TaMMA has been increasingly showing over the last months, we developed a similar meta-analysis of EoE-related public data sets visualized in an interactive web app, the EoE TaMMA, that includes studies analyzing EoE, GERD and controls (without EoE and GERD). EoE-related phenotypes were confirmed throughout the web app. To further consolidate the platform, we are proposing the validation of EoE TaMMA results in an independent cohort of EoE and GERD patients, by taking advantage of the EoE and GERD.

ELIGIBILITY:
Inclusion Criteria:

FFPE tissue samples patients who:

* had previously undergone endoscopic biopsy-collection in the clinical unit of Gastroenterology and Digestive Endoscopy according to the clinical practice (from 31/07/2012 to 31/07/2022)
* during that endoscopic biopsy-collection they already signed the attestation of will for using their clinical data for future scientific studies

Exclusion Criteria:

FFPE tissues from patients who:

- have not signed the attestation of will for authorized using the use of their clinical data for future scientific studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will use FFPE samples derived from patients who, at the time of the endoscopic exam, have signed the informed consent form to authorize the use of their clinical data for scientific purposes.
  We will validate the EoE TaMMA results (such as the upregulation of CCL26, TBX5, NOX4, FGF7, CXCL14, ADAMTS5, PDGFRA, CXCL12, ACVRL1, POSTN, and LTBP4 in EoE tissues by comparison with the GERD and the controls (without EoE and GERD)) by analyzing the EoE, GERD and controls FFPE samples already stored in the pathological laboratory.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the presence and the expression of several markers, including CCL26, TBX5, NOX4, FGF7, CXCL14, ADAMTS5, PDGFRA, CXCL12, ACVRL1, POSTN, and LTBP4 in FFPE tissue samples. | 1-12 months
  The investigators will use FFPE samples derived from patients who, at the time of the endoscopic exam, have signed the informed consent form to authorize the use of their clinical data for scientific purposes. The investigators will stain FFPE tissue samples with specific immunohistochemical antibodies, quantifying the presence of these specific markers: CCL26, TBX5, NOX4, FGF7, CXCL14, ADAMTS5, PDGFRA,CXCL12, ACVRL1, POSTN, and LTBP4.
  In order to perform the standard staining procedure, first the tissue section has to be deparaffinized and then rehydrated before applying the primary antibody. Enzyme-conjugated secondary antibodies are then applied, and the specific staining can be visualized after adding the enzyme- specific substrate.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided